CLINICAL TRIAL: NCT02228239
Title: A Double-blind, Randomized, Placebo-Controlled, 3-way Crossover Study to Evaluate the Single Dose Effects of Intranasal Esketamine on Safety of On-Road Driving in Healthy Subjects
Brief Title: Study to Assess the Effects of Esketamine on Safety of On-road Driving in Healthy Participants
Acronym: DRiVESaFe
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: CR104764; 2014-002005-38 (EudraCT Number); ESKETINTRD1006 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-08-27; First posted 2014-08-28 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
Keywords: Healthy; Esketamine; Mirtazapine; Psychomotor.
MeSH Terms: interventions — Esketamine; Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1 (ABC) (Experimental): Participants will receive Treatment A (esketamine 84 milligram (mg) intranasally and 1 placebo capsule) in Period 1, Treatment B (placebo intranasally and 1 mirtazapine 30 mg capsule) in Period 2 and Treatment C (placebo intranasally and placebo capsule) in Period 3 with a washout interval of at least 6 days between treatment periods.
  Interventions: Drug: Esketamine; Drug: Mirtazapine; Drug: Placebo (Matched to Esketamine); Drug: Placebo (Matched to Mirtazapine)
- Sequence 2 (BCA) (Experimental): Participants will receive Treatment B (placebo intranasally and 1 mirtazapine 30 mg capsule) in Period 1, Treatment C (placebo intranasally and placebo capsule) in Period 2 and Treatment A (esketamine 84 mg intranasally and 1 placebo capsule) in Period 3 with a washout interval of at least 6 days between treatment periods.
  Interventions: Drug: Esketamine; Drug: Mirtazapine; Drug: Placebo (Matched to Esketamine); Drug: Placebo (Matched to Mirtazapine)
- Sequence 3 (CAB) (Experimental): Participants will receive Treatment C (placebo intranasally and placebo capsule) in Period 1, Treatment A (esketamine 84 mg intranasally and 1 placebo capsule) in Period 2 and Treatment B (placebo intranasally and 1 mirtazapine 30 mg capsule) in Period 3 with a washout interval of at least 6 days between treatment periods.
  Interventions: Drug: Esketamine; Drug: Mirtazapine; Drug: Placebo (Matched to Esketamine); Drug: Placebo (Matched to Mirtazapine)
- Sequence 4 (CBA) (Experimental): Participants will receive Treatment C (placebo intranasally and placebo capsule) in Period 1, Treatment B (placebo intranasally and 1 mirtazapine 30 mg capsule) in Period 2 and Treatment A (esketamine 84 mg intranasally and 1 placebo capsule) in Period 3 with a washout interval of at least 6 days between treatment periods.
  Interventions: Drug: Esketamine; Drug: Mirtazapine; Drug: Placebo (Matched to Esketamine); Drug: Placebo (Matched to Mirtazapine)
- Sequence 5 (ACB) (Experimental): Participants will receive Treatment A (esketamine 84 mg intranasally and 1 placebo capsule) in Period 1, Treatment C (placebo intranasally and placebo capsule) in Period 2 and Treatment B (placebo intranasally and 1 mirtazapine 30 mg capsule) in Period 3 with a washout interval of at least 6 days between treatment periods.
  Interventions: Drug: Esketamine; Drug: Mirtazapine; Drug: Placebo (Matched to Esketamine); Drug: Placebo (Matched to Mirtazapine)
- Sequence 6 (BAC) (Experimental): Participants will receive Treatment B (placebo intranasally and 1 mirtazapine 30 mg capsule) in Period 1, Treatment A (esketamine 84 mg intranasally and 1 placebo capsule) in Period 2 and Treatment C (placebo intranasally and placebo capsule) in Period 3 with a washout interval of at least 6 days between treatment periods.
  Interventions: Drug: Esketamine; Drug: Mirtazapine; Drug: Placebo (Matched to Esketamine); Drug: Placebo (Matched to Mirtazapine)

INTERVENTIONS:
Drug: Esketamine — Esketamine 84 milligram (mg) [3*1 of spray in each nostril] will be administered intranasally on Day 1 in one of the treatment periods.
  Other Names: JNJ-54135419
Drug: Mirtazapine — Mirtazapine 30 mg capsule will be administered orally on Day 1 in one of the treatment periods.
Drug: Placebo (Matched to Esketamine) — Placebo [3*1 in each nostril] will be administered intranasally on Day 1 in one of the treatment periods.
Drug: Placebo (Matched to Mirtazapine) — Placebo capsule will be administered orally on Day 1 in one of the treatment periods.

SUMMARY:
The purpose of this study is to evaluate the effect of esketamine compared to placebo on driving performance as assessed by the mean difference of standard deviation of lateral position (SDLP) from an on-road driving test in healthy participants.

DETAILED DESCRIPTION:
This is a Phase 1, randomized (study medication assigned to participants by chance), double-blind (neither Investigator nor participant knows which treatment the participant receives), placebo-controlled (placebo is an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial), single-center, single-dose and 3-way crossover (the same medications provided to all participants but in different sequence) study of esketamine in healthy participants. Participants will be randomly assigned to 1 of 6 treatment sequences. The study will consist of 3 parts: Screening Phase (between 21 days and 1 day prior to the first dose administration), a 3-way crossover double-blind, single dose treatment Phase (45 days) and follow-up Phase (7 to 10 days after last dose administration). The maximum study duration for each participant will not exceed 7 weeks. Participants will receive either Treatment A (esketamine 84 milligram (mg) intranasal and 1 placebo capsule), Treatment B (placebo intranasal and 1 mirtazapine 30 mg capsule) or Treatment C (placebo intranasal and placebo capsule) in each treatment period. Driving performance will be assessed primarily by the mean difference of SDLP from an on road driving test. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) (weight [kg]/height^2[m^2]) between 18 and 30 kg/m^2 (inclusive), and body weight not less than 45 kg
* Blood pressure (after the participants is supine for 5 minutes) between 90 and 140 millimeter of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic at Screening and pre-dose on Day 1 of Period 1
* A woman of childbearing potential must have a negative urine pregnancy test at Screening and pre-dose on Day 1 of Period 1
* A 12-lead electrocardiogram (ECG) consistent with normal cardiac conduction and function at Screening and pre-dose on Day 1 of Period 1, including: sinus rhythm, heart rate between 45 and 90 beats per minute (bpm), QTc interval less than or equal to 450 milliseconds (ms), QRS interval of less than 120 ms, PR interval less than 200 ms and morphology consistent with healthy cardiac conduction and function 1st degree AV block is exclusionary
* Participant has a valid driving license for more than 3 years, has driven at least 5000 kilometer (km) in the past year and is driving a car regularly

Exclusion Criteria:

* Participant has clinically significant liver or renal insufficiency; cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic (including cataplexy and cognitive impairment), hematologic, rheumatologic, psychiatric, or metabolic disturbances. A significant primary sleep disorder is exclusionary
* Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at Screening, as deemed appropriate by the Investigator
* Clinically significant abnormal physical examination, vital signs, or 12-lead electrocardiogram (ECG) at Screening or on Day 1 of Period 1, as deemed appropriate by the Investigator
* Anatomical or medical conditions that may impede delivery or absorption of study medication (for example, undergone facial reconstruction, rhinoplasty, significant structural or functional abnormalities of the nose or upper airway; obstructions or mucosal lesions of the nostrils or nasal passages; undergone sinus surgery in the previous 2 years; or signs and symptoms of rhinitis predose on Day 1 of Period 1)
* Has an abnormal or deviated nasal septum with any one or more of the following symptoms: blockage of one or both nostrils, nasal congestion (especially 1-sided), frequent nosebleeds, frequent sinus infections, and at times has facial pain, headaches, and postnasal drip

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Standard Deviation of Lateral Position (SDLP) Assessed From an On-road Driving Test | 4 to 14 hours post-dose
  The SDLP will be measured from a validated on-road driving test in a 100 kilometer (km) highway-driving lane.

SECONDARY OUTCOMES:
Standard Deviation of Speed (SDS) Assessed From an On-road Driving Test | 4 to 14 hours post-dose
  The SDS will be measured from a validated on-road driving test in a 100 km highway-driving lane.
Mean Speed (MS) Assessed From an On-road Driving Test | 4 to 14 hours post-dose
  The MS will be measured from a validated on-road driving test in a 100 km highway-driving lane.
Mean Lateral Position (MLP) Assessed From an On-road Driving Test | 4 to 14 hours post-dose
  The MLP will be measured from a validated on-road driving test in a 100 km highway-driving lane.
Subjective Driving Performance Score | After completion of driving test (4 to 14 hours post-dose)
  Participants will indicate the perceived quality of their driving performance on a visual analog scale, which ranges from 0 ('I drove exceptionally poorly') to 20 ('I drove exceptionally well').
Karolinska Sleepiness Scale (KSS) Score | Pre-dose, 1, 2 hours and after completion of driving test (4 to 14 hours post-dose)
  The KSS is a participant-reported assessment used to rate sleepiness on a scale of 1 to 9, ranging from 1 (extremely alert) to 9 (very sleepy, great effort to keep awake, fighting sleep).
Columbia Suicide Severity Rating Scale (C-SSRS) Score | Up to 7 to 10 days after last dose administration
  The C-SSRS is a low-burden measure of the spectrum of suicidal ideation and behavior developed to assess severity and track suicidal events providing a summary of both suicidal ideation and behavior to identify the level and type of suicidality present.
Brief Psychiatric Rating Scale (BPRS) Symptom Sub-Scale Score | Pre-dose, 1 and 2 hours post-dose
  The BPRS is an 18-item rating scale which is used to assess a range of psychotic and affective symptoms rated from both observation of the participant and the participant's own report. Only the 4-item positive symptom subscale (consisting of: suspiciousness/persecution, hallucinations, unusual thought content, and conceptual disorganization) will be used and each question is rated on a 7-point scale ranging from 0 (not present) to 6 (extremely severe).
Clinician Administered Dissociative States Scale (CADSS) Score | Pre-dose, 1 and 2 hours post-dose
  The CADSS is an instrument for the measurement of present-state dissociative symptoms. The CADSS comprises 23 subjective items, divided into 3 components: Depersonalization, Derealization and Amnesia. Participant's responses are coded on a 5-point scale (0 = "Not at all" through to 4 = "Extremely").
Maximum plasma concentration (Cmax) | Pre-dose, 0.5, 1, 3 and 4 hours post-dose
  The Cmax is the maximum observed plasma concentration of esketamine or noresketamine.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Leiden, Netherlands